CLINICAL TRIAL: NCT02384915
Title: Spinale Unilaterale o Blocco Nervoso Periferico Per le Artroscopie di Ginocchio in Day Surgery. Confronto Prospettico Randomizzato
Brief Title: Spinal Anesthesia Versus Combined Sciatic-femoral Nerve Block for Outpatient Knee Arthroscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ASST Gaetano Pini-CTO (Other)
Responsible Party: Principal Investigator, Gianluca Cappelleri, Medical Doctor, ASST Gaetano Pini-CTO
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IOGPGC07
Record Dates: First submitted 2015-02-20; First posted 2015-03-10 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-03

CONDITIONS: Knee Arthritis
MeSH Terms: interventions — Prilocaine; Mepivacaine; Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spinal anesthesia (Experimental): Intrathecal injection of 2 ml (40 mg) of 2% hyperbaric prilocaine at L3-L4 interspaces through a 100mm Sprotte 25 G spinal needle (Pencan, b-brawn, Germay) in lateral decubitus position, (with limb to operate declive).
  Interventions: Drug: prilocaine; Procedure: Spinal anesthesia
- peripheral nerve block (Active Comparator): Ultrasound-guided sciatic-femoral nerve block injecting 25 ml of a 2% mepivacaine solution,15 ml on femoral nerve and 10 ml on sciatic nerve through a 80 mm 22g eco-reflex needle (Sonoplex, Pajunk, Germany)
  Interventions: Drug: mepivacaine; Procedure: Sciatic-femoral Nerve Block; Device: Sonoplex, Pajunk

INTERVENTIONS:
Drug: prilocaine
  Other Names: prilotekal
  Arms: Spinal anesthesia
Drug: mepivacaine
  Other Names: carbocaine
  Arms: peripheral nerve block
Procedure: Sciatic-femoral Nerve Block — ultrasound-guided 25 ml 2% mepivacaine injection on both femoral and sciatic nerve
  Arms: peripheral nerve block
Procedure: Spinal anesthesia — intrathecal injection of 40 mg hyperbaric prilocaine
  Arms: Spinal anesthesia
Device: Sonoplex, Pajunk
  Arms: peripheral nerve block

SUMMARY:
The aim of the study is to compare the time of home discharge in day-case patients receiving either a spinal anesthesia or a combined sciatic-femoral nerve block for knee arthroscopy

DETAILED DESCRIPTION:
Two groups: the first receive a spinal anesthesia injecting 2% hyperbaric prilocaine 40 mg with the patients in lateral decubitus and the surgical limb declive, the second a combined ultrasound-guided sciatic-femoral nerve block injecting 25 ml of 2% mepivacaine solution.

Onset time, performance time, duration of the block, time of voiding, as well as the time of home discharge will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* outpatients knee arthroscopy

Exclusion Criteria:

* diabetes
* allergy to local anesthetic
* patient refusal
* chronic opiods assumption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Time to home discharge | 12 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico G. Pini, Milan, Milano, Italy